CLINICAL TRIAL: NCT03869437
Title: Investigator Driven Randomized Controlled Trial of Cefiderocol Versus Standard Therapy for Healthcare Associated and Hospital Acquired Gram-negative Blood Stream Infection: Study Protocol (the GAME CHANGER Trial)
Brief Title: RCT Cefiderocol vs BAT for Treatment of Gram Negative BSI
Acronym: GAMECHANGER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAME CHANGER
Record Dates: First submitted 2019-02-06; First posted 2019-03-11 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Bloodstream Infections
MeSH Terms: conditions — Sepsis | interventions — Cefiderocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefiderocol (Experimental): Participants will receive Cefiderocol 2 grams administered intravenously over 3 hours, every 8 hours for a minium of 5 days and a maximun of 14 days.
  Interventions: Drug: Cefiderocol
- Best Available Therapy (BAT) (Active Comparator): BAT will be chosen by the investigator and intravenously administered per country-specific guidelines.
  Interventions: Other: Best Available Therapy

INTERVENTIONS:
Drug: Cefiderocol — 2 grams intravenously administered over 3 hours every 8 hours for a period of 5 to 14 days (dosage adjustment is necessary based on renal function).
  Other Names: S-649266
  Arms: Cefiderocol
Other: Best Available Therapy — Standard of care was determined by the investigator
  Arms: Best Available Therapy (BAT)

SUMMARY:
The purpose of this study is to determine whether a new antibiotic, Cefiderocol which works against a wide variety of gram negative bacteria, is equally effective as the antibiotics that are currently used as current standard of care.

DETAILED DESCRIPTION:
Infections with antibiotic resistant bacteria cause a significant burden of disease worldwide. Bloodstream infections may arise from a variety of sources, are commonly encountered in clinical practice, and are associated with significant morbidity and mortality. Antibiotics that have activity against a broad spectrum of pathogens are commonly suggested in treatment guidelines to adequately cover bloodstream infections. Increasing rates of resistance to antibiotics commonly used for bloodstream infection are problematic and may lead to initial empiric therapy not having activity against the pathogen isolated. In patients with bloodstream infections and sepsis, delay until the receipt of effective therapy is associated with an increase in mortality.

Increasing rates of antibiotic resistance in Gram-negative organisms due to the presence of extended spectrum beta lactamases (ESBL), hyperproduction of AmpC enzymes, carbapenemases and other mechanisms of resistance are identified in common hospital and healthcare associated pathogens including Enterobacteriaceae, Pseudomonas aeruginosa and Acinetobacter baumannii. Uncommonly, Gram-negative organisms such as Klebsiella pneumoniae and, in tropical areas such as south-east Asia and northern Australia, Burkholderia pseudomallei can cause severe community-acquired pneumonia resulting in bloodstream infection.

Cefiderocol (previously S-649266) is a novel siderophore cephalosporin antibiotic with a catechol moiety on the 3-position side chain. The catechol side chain enables ferric iron ion binding, and the resulting complex of cefiderocol and iron ions is actively transported into bacteria via ferric iron transporter systems with subsequent destruction of cell wall synthesis. Cefiderocol has been shown to be potent in vitro against a broad range of Gram-negative organisms, including carbapenem-resistant Enterobacteriaceae (CRE) and multi-drug resistant (MDR) P. aeruginosa and A. baumannii . This activity is considered to be due to not only efficient uptake via the active siderophore systems but also the high stability of cefiderocol against carbapenemase hydrolysis. Limited in vitro data suggests cefiderocol may have activity against B. pseudomallei.

Recent clinical data has shown cefiderocol to be effective in the setting of complicated urinary tract infections , including patients with concomitant bacteremia. A study examining the use of cefiderocol in the setting of infections caused by carbapenem-resistant organisms is currently underway, as is a study of cefiderocol for hospital acquired pneumonia (ClinicalTrials.gov NCT02714595 & NCT03032380). Given the broad spectrum of activity against Gram-negative organisms, including those with resistant phenotypes, cefiderocol may be an ideal agent for empiric use in the setting of bloodstream infections acquired in the hospital or healthcare setting but as yet no clinical trial has examined this.

ELIGIBILITY:
Inclusion Criteria:

1. Bloodstream infection with a Gram-negative organism from at least one blood culture draw. Bacterial identification to species level will be performed using standard laboratory methods (e.g. MALDI-TOF) and susceptibility testing (e.g. Vitek2).
2. The blood stream infection fulfils the criteria as a hospital acquired or healthcare associated infection as per the following definitions:

   1. Hospital acquired - Blood stream infection occurring greater than 48 hours after hospital admission, assessed as symptoms or signs of infection not present at time of hospital admission.
   2. Healthcare associated - Blood stream infection present at admission to hospital or within 48 hours of admission in patients that fulfil ANY of following criteria:

   i. Participant has an intravascular catheter/line that is the source of infection ii. Attended a hospital or haemodialysis clinic or received intravenous chemotherapy in the previous 30 days iii. were hospitalized in an acute care hospital for two or more days in the previous 90 days iv. resided in a nursing home or long-term care facility v. received intravenous antibiotic therapy at home, wound care or specialized nursing care through a healthcare agency, family or friends; or had self-administered intravenous antibiotic medical therapy in the 30 days before the infection
3. No more than 48 hours has elapsed since the positive blood culture collection.
4. Participant is aged 18 years and over (21 in Singapore)
5. The participant or approved proxy is able to provide informed consent.

Exclusion Criteria:

1. Refractory shock or comorbid condition such that patient not expected to survive more than 7 days.
2. Participant with history of moderate to severe hypersensitivity reaction to a cephalosporin.
3. Participant with significant polymicrobial bacteraemia including a significant Gram-positive pathogen (that is, a Gram-positive skin contaminant in one set of blood cultures is not regarded as significant polymicrobial bacteraemia).
4. Where the bloodstream infection is thought to be related to a vascular catheter and the catheter is unable to be removed.
5. Treatment is not with the intent to cure the infection (that is, palliative care is an exclusion).
6. Known pregnancy or breast-feeding.
7. Participant is receiving peritoneal dialysis.
8. Participant previously randomised in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Mortality at 14 days | 14 days post date of randomisation
  To compare the 14-day mortality from day of randomisation of each regimen (cefiderocol versus standard of care therapy). If the primary objective meets the criteria for non-inferiority (with a margin of 10% for the difference in proportions), superiority will be examined.

SECONDARY OUTCOMES:
Mortality post blood stream infection of each regimen at longer time points | 30 and 90 days, from day of randomisation or "day 1"
  If a date of death is recorded on or before our calculation of Day 14, the participant will be classed as dead, otherwise considered to be alive. Similar for Day 30. Where possible this rule will also be applied for Day 90 vital status. If the Day 90 follow-up actually occurred on day 85 to 89 and the participant was alive we will assume the participant was alive at day 90.
Clinical and microbiological failure at day 14 | Day 14, from day of randomisation or "day 1"
  Defined as composite of:
  1. Death
  2. Still in hospital and clinical failure, as deﬁned by
     1. If baseline SOFA ≥3, D(day)14 SOFA not improved by ≥30%
     2. If baseline SOFA <3, D14 SOFA worse
  3. Microbiological failure (GNB Growth in blood of same species as index GNB from days 3-14)
  The SOFA score we will calculate is a slight modiﬁcation of the original SOFA score. It will be used for ICU and non-ICU participants. The sole modiﬁcation is that the respiratory component will be scored as in the modiﬁed SOFA:
  * 0 (if SaO2/FiO2 >400)
  * 1 (if SaO2/FiO2 315-400)
  * 2 (if SaO2/FiO2 235-314)
  * 3 (if SaO2/FiO2 150-234)
  * 4 (if SaO2/FiO2 <150)
Microbiological failure days 3 to 90 post randomisation | Day 3 through to day 90
  Deﬁned as growth in blood cultures of the same GNB as the index blood culture(s), from day 3 up to day 90.
Colonisation or infection with methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant enterococci (VRE), carbapenem-resistant Gram-negative bacilli or Candida bloodstream infection. | Day 3 through to day 90
  Deﬁned as the presence of MRSA, VRE or carbapenem-resistant Gram-negative bacilli (of a diﬀerent species from primary BSI organism) on culture +/- molecular test of clinical samples or screening swabs, or Candida species grown in blood cultures from day 3 up to day 90.
Clostridioides diﬃcile infection days 3 to 90 post randomisation. | Day 3 through to day 90
  Deﬁned as presence of a compatible clinical illness with a positive laboratory stool test for C. diﬃcile (as per local diagnostic protocol / method).
Improvement in functional status at day 30 post randomisation compared to baseline. | Day 30, from day of randomisation or "day 1"
  Functional status will be measured according to a score ranging from 0 (dead) to 7 (out of hospital, healthy, able to complete daily actvities). This score is based on the Functional Bloodstream Infection Score (FBIS) [McNamara et al. Clin Microbiol Infect. 2020 Feb;26(2):257.e1-257].
Time to hospital discharge. | From day of randomisation or "day 1" through to day 90
  Deﬁned as to the day of ﬁrst discharge alive (e.g. Day 2 is the day after randomisation). However, if a participant dies in the 3 days following ﬁrst hospital discharge, we will consider that participant as not having a discharge alive.
Treatment emergent SAEs (Serious Adverse Events) | From day of randomisation or "day 1" through to 5 days post end of study treatment.
  Defined as a serious adverse event possibly, probably or definitely related to the randomised drug treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Paterson, Professor, Principal Investigator — The Univeristy of Queensland
Locations (19):
- Australia (5):
  - Westmead Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Brisbane and Womens Hospital, Brisbane, Queensland
  - The Prince Charles Hospital, Brisbane, Queensland
  - Austin Hospital, Melbourne, Victoria
- Malaysia (2):
  - Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - University of Malaya Medical Centre, Kuala Lumpur
- Singapore (4):
  - Changi General Hospital, Singapore
  - National University Hospital Singapore, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Thailand (3):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Khon Kaen University, Khon Kaen
- Istanbul Medipol Üniversitesi, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Paterson DL, Sulaiman H, Liu PY, Chatfield MD, Yilmaz M, Salmuna ZN, Mazlan MZ, Anunnatsiri S, Sirijatuphat R, Chotiprasitsakul D, Lye DC, Somani J, Kalimuddin S, Aslan AT, Thamlikitkul V, Lee YT, Yang YS, Lin YT, Ramli WNW, Tseng CH, Archuleta S, Chan YFZ, Forde BM, Wright H, Stewart AG, Ramsay KA, Ling W, Rossi V, Harris-Brown TM, Harris PNA; GAME CHANGER Trial Investigators. Cefiderocol versus standard therapy for hospital-acquired and health-care-associated Gram-negative bacterial bloodstream infection (the GAME CHANGER trial): an open-label, parallel-group, randomised trial. Lancet Infect Dis. 2026 Feb;26(2):148-159. doi: 10.1016/S1473-3099(25)00469-4. Epub 2025 Oct 6. PMID 41067237
- [Derived] Wright H, Harris PNA, Chatfield MD, Lye D, Henderson A, Harris-Brown T, Donaldson A, Paterson DL. Investigator-Driven Randomised Controlled Trial of Cefiderocol versus Standard Therapy for Healthcare-Associated and Hospital-Acquired Gram-negative Bloodstream Infection: Study protocol (the GAME CHANGER trial): study protocol for an open-label, randomised controlled trial. Trials. 2021 Dec 7;22(1):889. doi: 10.1186/s13063-021-05870-w. PMID 34876196

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT03869437/SAP_000.pdf